CLINICAL TRIAL: NCT03493230
Title: Detection of Plasmatic Cell-free BRAF and NRAS Mutations: a New Tool for Monitoring Patients with Metastatic Malignant Melanoma Treated with Targeted Therapies or Immunotherapy ( MALT )
Brief Title: Detection of Plasmatic Cell-free BRAF and NRAS Mutations : a New Tool for Monitoring Patients with Metastatic Malignant Melanoma Treated with Targeted Therapies or Immunotherapy ( MALT )
Acronym: MALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-AOI-07
Record Dates: First submitted 2018-03-26; First posted 2018-04-10 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Malignant Melanoma Stage IV; Malignant Melanoma Stage III
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with malignant melanoma (Experimental): Patient with advanced or metastatic malignant melanoma (stage IIIB inoperable or IIIC or stage IV) will have a first blood test before any treatment, then at day 15 or 30 after initiation of therapy, and every two months until recurrence or progression for a maximum of 22 months.
  Interventions: Biological: quantification of BRAF and NRAS mutation

INTERVENTIONS:
Biological: quantification of BRAF and NRAS mutation — Quantification of cell-free BRAF and NRAS mutations with digital PCR

SUMMARY:
The main objective of this project is to perform a longitudinal monitoring of BRAF and NRAS cell-free DNA in a large cohort of metastatic melanomas patients before treatment and during the follow-up. Results will be compared with clinical data as imaging (based on RECIST criteria) and the activity of lactate dehydrogenase in serum (LDH).

DETAILED DESCRIPTION:
During a consultation of follow-up for an advanced malignant melanoma (stage IIIb or IIIC or IV), an investigator presents the study to the patient and give him the note of information and the informed consent.

The patient can benefit from a reflexion period of of 7 days.

In case of agreement, a first blood draw will take place before initiation of any treatment. Between D15 and D30 a second blood draw will be taken. Then a blood draw will be necessary every two months until recurrence or progression of the disease for a maximum of 22 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients in metastatic situation for a malignant melanoma inoperable stage IIIB or IIIC or stage IV
* In first line of treatment by a targeted therapy (only or in association) or immunotherapy
* Every histological types of cutaneous or mucous malignant melanoma (excepted choroid melanomas)
* The tumor must be mutates for BRAF or NRAS
* The mutation status must have been realized in the Laboratory Pathology Clinical and Experimental (LPCE) of the CHU de Nice analysis of the status on-site metastatic mutational and/or primitive tumor must
* Membership or beneficiary of the national insurance scheme

Exclusion Criteria:

* Histories of cancer or other synchronous cancer
* Pregnant, breast-feeding Women. A pregnancy test will be practiced to the women old enough to procreate.
* Vulnerable People: adults under guardianship, patients deprived of freedom, minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Quantify plasmatic BRAF and NRAS mutation determine by PCR digitale in µg/ml before treatment | Day 0
Study the longitudinal monitoring of cell-free the kinetics of the plasma mutation of BRAF and NRAS mutation in µg/ml and comparing them with imaging (based on RECIST criteria) and with the activity of the lactate dehydrogenase in serum ( LDH) in U/l . | Month 24

SECONDARY OUTCOMES:
Compare the results obtained by PCR digitale from the cell-free with the results on FFPE tissue samples | Month 24
Identify genomic alterations and mutations of resistances in a restricted subgroup of patient by New Generation Sequencing analysis | Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Elodie LONG-MIRA, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- nice University hospital, Nice, France

REFERENCES:
- [Background] Bahadoran P, Allegra M, Le Duff F, Long-Mira E, Hofman P, Giacchero D, Passeron T, Lacour JP, Ballotti R. Major clinical response to a BRAF inhibitor in a patient with a BRAF L597R-mutated melanoma. J Clin Oncol. 2013 Jul 1;31(19):e324-6. doi: 10.1200/JCO.2012.46.1061. Epub 2013 May 28. No abstract available. PMID 23715574
- [Background] de Vries E, Bray FI, Coebergh JW, Parkin DM. Changing epidemiology of malignant cutaneous melanoma in Europe 1953-1997: rising trends in incidence and mortality but recent stabilizations in western Europe and decreases in Scandinavia. Int J Cancer. 2003 Oct 20;107(1):119-26. doi: 10.1002/ijc.11360. PMID 12925966
- [Background] Dhillon AS, Hagan S, Rath O, Kolch W. MAP kinase signalling pathways in cancer. Oncogene. 2007 May 14;26(22):3279-90. doi: 10.1038/sj.onc.1210421. PMID 17496922